CLINICAL TRIAL: NCT02287116
Title: Continuous Positive Airway Pressure Via Binasal Prong vs Nasal Mask: a Randomised Controlled Trial
Acronym: MASK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Principal Investigator, birgul say, CONTINUOUS POSITIVE AIRWAY PRESSURE VIA BINASAL PRONG VS NASAL MASK: A RANDOMISED CONTROLLED TRIAL, Zekai Tahir Burak Women's Health Research and Education Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BIRBILYA; BS197455 (Other Grant/Funding Number: BS197455)
Record Dates: First submitted 2014-11-02; First posted 2014-11-10 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Bronchopulmonary Dysplasia; Death
Keywords: preterm infants; CPAP; BPD; invasive mechanical ventilation; we aimed determine that affect the rate of BPD and death of NCPAP therapy with nasal prongs or nasal mask as the initial treatment for RDS.
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Death

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- nasal mask and nasal prongs (No Intervention)
  Interventions: Device: Easy Flow system and INCA® nasal cannulae set

INTERVENTIONS:
Device: Easy Flow system and INCA® nasal cannulae set

SUMMARY:
The investigators aimed to compare the effectiveness of nasal mask and prongs used in CPAP (nasal continuous positive airway pressure)as the initial respiratory support when using minimal ly invasive surfactant therapy (MIST) in preterm infants.

DETAILED DESCRIPTION:
OBJECTIVE: To determine that affect the rate of (bronchopulmonary dysplasia) BPD and death of NCPAP therapy with nasal prongs or nasal mask as the initial treatment for respiratory distress syndrome (RDS).

METHODS: Inborn preterm infants of gestational age 26-32 weeks, with respiratory distress syndrome were enrolled in this single-centered, unblinded randomized prospective controlled trial. They were stabilized with T-piece device in delivery room. Immediately after admission of neonatal intensive care unit (NICU), infants were randomly assigned to receive NCPAP with either nasal prongs or mask. NCPAP was continued by setting at PEEP as 5 to 8 cm H2O .

RESULTS: 160 infants were assessed for eligibility 149 infants were randomized. Finally 75 infants in Group I (nasal prong) and 74 in Group II (nasal mask) were analyzed. Mean gestational ages were 29.3±1.6 vs 29.1±2.0 weeks (p=0.55) and birth weights were 1225±257 vs. 1282±312 grams (p=0.22) respectively in Group I and Group II. The frequency of NCPAP failure within 24 hours of life was higher in Group I compared to Group 2 (respectively 8%, %0 , p=0.09) but difference was not significant. The outcomes of BPD and death rates did not differ among the groups ( Group I 9.3% vs. Group II 9.4 %; p=0.96).

CONCLUSIONS: Applied nasal mask is a feasible method to deliver NCPAP and as effective as nasal prongs for the initial treatment of RDS in preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* One hundred sixty infants born at 26-32 weeks' gestation not endotracheally intubated in the delivery room (DR)

Exclusion Criteria:

* Infants with major congenital anomalies, and who required intubation in the DR and no parental consent were excluded.

Max Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2014-05; Primary Completion 2014-05 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
BPD | 7 months
  To determine that affect the rate of BPD of NCPAP therapy with nasal prongs or nasal mask as the initial treatment for RDS.

SECONDARY OUTCOMES:
death | 7
  To determine that affect the rate of death of NCPAP therapy with nasal prongs or nasal mask as the initial treatment for RDS.